CLINICAL TRIAL: NCT01198678
Title: Feasibility Study to Assess the Safety and Functionality of the GluSense-LTone 2e3 Continuous Glucose Monitor in Diabetic Patients
Brief Title: Feasibility Study to Assess the Safety and Functionality of the GluSense Continuous Glucose Monitor in Diabetic Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GluSense Ltd (Industry)
Responsible Party: Dr. Tehila Hyman, GluSense Ltd
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: Slovenia-UMC-001
Record Dates: First submitted 2010-09-08; First posted 2010-09-10 (Estimated); Last update posted 2011-03-31 (Estimated); Status verified 2010-12

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: Boost Nutritional Supplement — Boost- Nutritional Supplement
  Other Names: boost HP

SUMMARY:
Currently marketed CGM sensors have an approved functional lifetime of up to 1 week. Pre-clinical studies have demonstrated that GluSense-LTone 2e3 sensors may be used to accurately monitor glucose levels for 30 days. The purpose of this study is to assess the safety and functionality of the device in human patients for consecutive 15 days.

GluSense-LTone 2e3 as long term CGM, will require less sensor replacements and calibration, meaning less patient interventions, and is therefore will be much more user friendly. Moreover, GluSense-LTone 2e3 shows potentially increased accuracy, especially in the critically important hypoglycemic range, meaning that better management of patient's condition may be attained.

DETAILED DESCRIPTION:
GluSense-LTone 2e3 is a continuous glucose monitoring (CGM) system. It is a semi-invasive, optical fiber-based device with a lifetime of up to one month. The purpose of this study is to assess the safety, accuracy, calibration requirements and effective lifetime of the device.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be eligible for participation in this study:

* Male or female patients between 18 and 50 years of age
* Patients with type 1 diabetes mellitus.
* The ability to read, understand and sign an informed consent form. Written consent must be obtained prior to initiation of study procedures

Exclusion Criteria:

Patients who meet any of the following exclusion criteria are not to be enrolled in this study:

* Clinical significant illness that can compromise patient's health during study such as:

  * Significant current heart disease
  * Significant Liver or kidney disease
  * HIV infection
  * Hepatitis B or Hepatitis C infection
  * Malignancy
  * Major allergic skin disease including plaster allergies
  * Significant allergic disorders
* Current or recent significant skin conditions (e.g. eczema, psoriasis,).
* Presence of skin markings/ abnormalities around implantation site that will interfere with the skin assessment e.g. tattoos, piercings, birthmark, sunburn
* Current alcohol or substance use judged by the IP to potentially interfere with patient study compliance.
* Routine administration of Steroid based medications.
* Patients currently taking part in any other clinical trial using an investigational product within the last 3 months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2010-11; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Evaluate capability to follow glucose concentration changes over 15 consecutive days | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tadej Batellino, Prof, Principal Investigator — University Medical Centre Ljubljana
Locations (1):
- University medical Center Ljubljana, Ljubljana, Slovenia